CLINICAL TRIAL: NCT07349888
Title: Combined Mitral and Tricuspid Versus Isolated Mitral Transcatheter Edge-to-Edge Repair for Mitral Regurgitation With Tricuspid Regurgitation: A Randomized Controlled Trial
Brief Title: Combined Mitral and Tricuspid Versus Isolated Mitral Transcatheter Edge-to-Edge Repair for Mitral Regurgitation With Tricuspid Regurgitation (DUAL-TEER Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20251223-08
Record Dates: First submitted 2026-01-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Mitral Regurgitation; Tricuspid Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Tricuspid Valve Insufficiency | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Mitral and Tricuspid TEER (Experimental): Participants undergo simultaneous transcatheter edge-to-edge repair for mitral regurgitation and tricuspid regurgitation, accompanied by guideline-directed medical therapy (GDMT)
  Interventions: Device: Transcatheter Edge-to-Edge Repair (TEER) System
- Mitral TEER (Active Comparator): Participants undergo isolated mitral transcatheter edge-to-edge repair for mitral regurgitation, accompanied by GDMT
  Interventions: Device: Transcatheter Edge-to-Edge Repair (TEER) System

INTERVENTIONS:
Device: Transcatheter Edge-to-Edge Repair (TEER) System — Participants assigned to this arm will undergo simultaneous transcatheter edge-to-edge repair (TEER) for mitral and/or tricuspid regurgitation. All participants will receive guideline-directed medical therapy (GDMT) for heart failure and valvular heart disease throughout the study period.

SUMMARY:
This study aims to investigate the efficacy and safety of combined mitral and tricuspid transcatheter edge-to-edge repair (TEER) versus isolated mitral TEER in the treatment of patients with mitral regurgitation (MR) combined with tricuspid regurgitation (TR). The expected objective is to provide a more precise treatment strategy for patients with MR combined with TR, reduce surgical risks, improve survival rates and quality of life, and offer evidence for clinical practice. The main research content involves enrolling 404 patients with severe MR combined with TR, who will be randomly assigned to either the group receiving simultaneous mitral and tricuspid TEER or the group receiving isolated mitral TEER. The primary endpoint is the composite endpoint at one year postoperatively, including death during the one-year follow-up, mitral and/or tricuspid surgery or intervention due to mitral and/or tricuspid dysfunction, rehospitalization for heart failure, and an increase of <15 points in the KCCQ score.

ELIGIBILITY:
Inclusion Criteria General Inclusion Criteria

* Age ≥ 18 years
* Moderate-to-severe or severe (≥3+) degenerative mitral regurgitation (DMR) or functional mitral regurgitation (FMR) combined with severe (≥3+) functional tricuspid regurgitation (FTR)
* New York Heart Association (NYHA) functional class II, III, or IVa
* Anatomically suitable for transcatheter edge-to-edge repair, as assessed by the Heart Team
* Willing and able to comply with the protocol requirements and data collection procedures
* Capable of understanding the purpose of the trial and voluntarily providing written informed consent, either personally or via a legally authorized representative DMR Inclusion Criteria
* Symptomatic moderate-to-severe or severe degenerative mitral regurgitation (MR ≥3+)
* High surgical risk FMR Inclusion Criteria
* Symptomatic moderate-to-severe or severe functional mitral regurgitation (MR ≥3+)

For ventricular FMR:

* Left ventricular ejection fraction (LVEF) < 50%
* Persistent symptoms despite optimized guideline-directed medical therapy (GDMT) and cardiac resynchronization therapy (CRT), if indicated
* Clinically stable for at least 30 days prior to enrollment

For atrial FMR:

* Unsuitable for surgery
* Persistent symptoms despite optimized medical therapy
* Clinically stable for at least 30 days prior to enrollment TR Inclusion Criteria
* Severe functional tricuspid regurgitation (TR ≥3+)
* Persistent symptoms despite guideline-directed medical therapy (GDMT)
* Clinically stable for at least 30 days prior to enrollment

Exclusion Criteria:

* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or other structural heart disease causing heart failure (except dilated cardiomyopathy of ischemic or non-ischemic etiology)
* Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
* Refractory heart failure requiring advanced therapies (e.g., left ventricular assist device or heart transplantation)
* Left ventricular end-systolic diameter (LVESD) > 70 mm
* Left ventricular ejection fraction (LVEF) ≤ 20%
* Pulmonary arterial hypertension as assessed by right heart catheterization (RHC)
* Severe right ventricular dysfunction, defined as:

Tricuspid annular plane systolic excursion (TAPSE) < 10 mm, or Right ventricular tissue Doppler imaging S' < 6 cm/s, or Fractional area change (FAC) ≤ 22%

-Hemodynamic instability, defined as: Systolic blood pressure < 90 mmHg with afterload reduction, or Cardiogenic shock requiring inotropic support, intra-aortic balloon pump, or ther mechanical circulatory support

* Severe uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg)
* Myocardial infarction or unstable angina within 30 days prior to enrollment
* Significant untreated coronary artery disease requiring revascularization, or coronary intervention performed within 30 days prior to enrollment
* Moderate or greater aortic valve or pulmonary valve stenosis or regurgitation Mitral valve anatomy deemed unfavorable for transcatheter edge-to-edge repair by the Heart Team, including:Moderate-to-severe calcification in the grasping zone; Mitral valve orifice area < 3.5 cm²; Posterior mitral leaflet length < 7 mm; Mitral stenosis; Leaflet perforation; Multi-segment disease or multiple chordal rupture Tricuspid valve anatomy deemed unfavorable for transcatheter edge-to-edge repair by the Heart Team, including:Moderate-to-severe calcification in the grasping zone; Coaptation gap ≥ 10 mm; Severe leaflet perforation, cleft lesions, or other conditions preventing device implantation
* Congenital Ebstein's anomaly
* Prior surgical or interventional procedure involving the mitral or tricuspid valve
* Pacemaker or implantable cardioverter-defibrillator (ICD) leads interfering with proper device positioning
* Intracardiac thrombus, vegetation, mass, or tumor in the atria or ventricles
* Cerebrovascular accident (stroke) within 3 months prior to enrollment
* Chronic obstructive pulmonary disease requiring continuous home oxygen therapy or long-term outpatient oral steroid treatment
* End-stage renal disease requiring chronic dialysis
* Vascular access limitations, including inferior vena cava filter, severely tortuous or obstructed caval system, or difficult transseptal puncture
* Contraindications to antithrombotic therapy, or history of intracerebral hemorrhage, gastrointestinal bleeding, or bleeding disorders within 3 months prior to enrollment
* Uncontrolled active infection, including active bacterial endocarditis
* Severe comorbidities that may complicate treatment evaluation (e.g., coma, malignancy, or severe psychiatric disorders)
* Pregnancy or breastfeeding
* Life expectancy < 1 year
* Participation in another clinical trial that has not yet reached its primary endpoint
* Investigator judgment that the patient is non-compliant or unlikely to complete follow-up as required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint at 12 months | 12 months
  Including all-cause mortality, mitral and/or tricuspid valve surgery or intervention due to mitral and/or tricuspid valve dysfunction, heart failure rehospitalization, and a KCCQ score improvement of less than 15 points.

SECONDARY OUTCOMES:
All-cause mortality | Perioperative, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  all-cause mortality
Cardiovascular mortality | Perioperative, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Cardiovascular mortality
Incidence of surgical procedures due to mitral and/or tricuspid valve dysfunction | Perioperative, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Incidence of surgical procedures due to mitral and/or tricuspid valve dysfunction
Incidence of interventional procedures due to mitral and/or tricuspid valve dysfunction | Perioperative, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Incidence of interventional procedures due to mitral and/or tricuspid valve dysfunction
Incidence of heart failure rehospitalization | Perioperative, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Incidence of heart failure rehospitalization
Cardiac function change | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Change in New York Heart Association (NYHA) Functional Classification, a clinician-assessed scale ranging from Class I to Class IV, with higher class indicating worse functional status.
Quality of life of patients | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score, a patient-reported outcome measure ranging from 0 to 100, with higher scores indicating better health-related quality of life.
Quality of life of patients | Perioperative, 6 months, 12 months
  Changes in 6-minute walking distance
Technical success | Perioperative
  Successful implantation of the transcatheter edge-to-edge repair system, with immediate postoperative echocardiographic assessment showing MR and/or TR ≤2+, and no death or surgical reintervention prior to discharge.
The incidence of major adverse cardiovascular and cerebrovascular events during the trial (MACCEs) | Perioperative, 30 days, 6 months, 12 months
  Cardiac death, stroke, myocardial infarction, renal disease requiring unplanned dialysis or renal replacement therapy, unplanned or urgent intervention (interventional or surgical procedure) due to device-related complications, severe bleeding (as defined by MVARC), and access-related vascular complications requiring intervention.